CLINICAL TRIAL: NCT06791187
Title: The Effect of a Single Dose of BI 1291583 on the Pharmacokinetics of a Single Dose of Dabigatran Following Oral Administration in Healthy Adult Male Subjects (an Open-label, 2- Period, Fixed-sequence Study)
Brief Title: A Study in Healthy People to Test Whether BI 1291583 Influences the Amount of Dabigatran in the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1397-0022; 2024-516256-18-00 (Registry Identifier: CTIS); U1111-1312-4162 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-01-20; First posted 2025-01-24 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran

STUDY DESIGN:
Intervention Model Description: Participants cross over from test treatment (T) to reference treatment (R) (two periods, fixed sequence).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dabigatran alone (R) followed by dabigatran + BI 1291583 combination (T) (Experimental): R=reference treatment (period 1) T=test treatment (period 2)
  Interventions: Drug: dabigatran etexilate; Drug: BI 1291583

INTERVENTIONS:
Drug: dabigatran etexilate — dabigatran etexilate
  Other Names: Pradaxa
Drug: BI 1291583 — BI 1291583
  Other Names: Verducatib

SUMMARY:
The main objective of this trial is to investigate the effect of a single dose of BI 1291583 on the pharmacokinetics of a single dose of dabigatran, an efflux transporter P-glycoprotein (P-gp) substrate.

ELIGIBILITY:
Inclusion Criteria :

Subjects will only be included in the trial if they meet the following criteria:

1. Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 55 years (inclusive)
3. Body Mass Index (BMI) of 18.5 to 29.9 kg/m 2 (inclusive)
4. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial

Exclusion Criteria :

Subjects will not be allowed to participate, if any of the following general criteria apply:

1. Any finding in the medical examination (including Blood pressure (BP) Pulse rate (PR) or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
8. History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2025-01-23 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of dabigatran in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | Up to 4 days
Maximum measured concentration of dabigatran in plasma (Cmax) | Up to 4 days

SECONDARY OUTCOMES:
Area under the concentration-time curve of dabigatran in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com